CLINICAL TRIAL: NCT03077061
Title: Reconstructive Surgical Therapy of Peri-implantitis-related Osseous Defects. A Multicenter Randomized Controlled Clinical Trial
Brief Title: Peri-implantitis - Reconstructive Surgical Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1192-16
Record Dates: First submitted 2017-02-24; First posted 2017-03-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: The study is designed as a two-arm randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Individuals assessing radiographic parameters will be masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Open flap debridement (Active Comparator): The surgical procedure includes flap elevation, debridement of the peri-implant defect and decontamination of the implant surfaces using saline for irrigation. Flaps are replaced in their original position and carefully sutured. Patients are provided with post-surgical information and thereafter called in for regular follow-up visits.
  Interventions: Procedure: Open flap debridement
- Test - Bone replacement graft (Experimental): The surgical procedure is identical to the control procedure with the exception of the application of the bone replacement graft. Following decontamination, Bio-Oss Collagen® is placed into the peri-implant bony defect. Flaps are carefully sutured and patients are provided with the same information and follow-up as patients in the control group.
  Interventions: Procedure: Open flap debridement; Device: Bone replacement graft

INTERVENTIONS:
Procedure: Open flap debridement — Open flap debridement using saline as irrigation
Device: Bone replacement graft — Open flap debridement using saline as irrigation including a grafting procedure withBio-Oss Collagen®.
  Other Names: Bio-Oss Collagen®
  Arms: Test - Bone replacement graft

SUMMARY:
The project will evaluate the potential benefit of the use of bone replacement graft as an adjunct to surgical therapy of peri-implantitis. The project will be conducted as a two-armed randomized controlled clinical trial of 5-year duration in 7 clinical centers. 140 systemically healthy patients diagnosed with peri-implantitis will randomly assigned to be treated with or without bone replacement graft. Outcome measures include assessments of inflammation, probing depth, recession, radiological parameters and PROMs.

DETAILED DESCRIPTION:
Objective The overall objective of the project is to evaluate the clinical efficacy of the use of a bone substitute material in reconstructive surgical therapy of peri-implantitis-associated osseous defects.

Hypothesis: The use of a bone substitute material in reconstructive therapy of peri-implantitis increases the likelihood to achieve treatment success.

Relevance for clinical practice The project will provide significant contribution to the understanding of outcomes using reconstructive procedures in treatment of peri-implantitis.

Study population, design and treatment procedures The project will be conducted as a two-armed randomized controlled clinical trial of 5-year duration in 7 clinical centers. 140 systemically healthy patients with implants ≥1 year in function and diagnosed with advanced peri-implantitis at ≥1 implants will be enrolled.

Inclusion criteria Age ≥ 18 years

≥1 implant (≥1 year of function) presenting with PPD ≥7 mm and BoP/Pus. Confirmed bone loss ≥3 mm at same implant(s)

Exclusion criteria Treated for peri-implantitis during previous 6 months Intake of systemic or local antibiotics during previous 6 months Systemic conditions affecting peri-implant tissues Systemic conditions impeding surgical intervention

Surgical procedures Surgical procedures will be performed one month after a baseline examination and initiation of plaque control. Three days before surgery a 10-day systemic antibiotic regimen will be initiated. Full thickness flaps will be elevated and inflamed tissues will be removed. The implant surfaces will be cleaned with mini-gauze soaked in saline. The osseous defect should be ≤4 mm wide and >3 mm deep. The defect should in addition to the mesial and distal bone walls preferably exhibit at least a lingual or a buccal bone wall. The randomly assigned treatment strategy, stratified for smoking, will be revealed after debridement. Test procedure: The defect will be filled with Bio-Oss Collagen® and the flaps will be sutured to their previous position. Control procedure: Flaps will be sutured to their previous position. Sutures will be removed 2 weeks after treatment, followed by a 6-week control. Clinical examinations will be performed at 6, 12, 24, 36, 48 and 60 months after therapy. Maintenance therapy will be provided based on individual needs.

Clinical assessments One calibrated examiner in each clinical center will perform the assessments. The following variables will be assessed at four sites around the implant: Plaque, probing pocket depth (PPD), bleeding on probing (BoP), probing attachment level (PAL) and recession (REC).

Treatment success Treatment success will be defined as the absence of BoP/Pus, PPD ≤5 mm and ≤1 mm recession. Peri-implant sites showing BoP and PPD ≥6 mm at re-examination will be scheduled for further treatment. Patient-related outcome variables will be assessed at baseline and follow-up and include esthetic and functional appreciation, pain or discomfort.

Radiographic assessments Intra-oral radiographs will be obtained prior to surgery (baseline) and at 1-, 3- and 5-year re-examinations. Analysis of radiographs will be performed by specialists in oral-maxillofacial radiology. The examiners will be blinded to treatment procedures. The assessment will include defect fill and crestal bone support.

Power calculation A total of 122 patients (61 per group) will provide a power of 80% with alpha set at 0.05 to detect a difference of 1 mm in mean PPD change between groups, given a SD of 1.97 (Carcuac et al., 2016). 140 individuals will be included to compensate for drop-out.

Data analysis Mean changes for the various variables and the proportion of sites fulfilling the criteria for treatment success will be calculated. A multilevel model with the clinical center as the highest level and the implant as the lowest will be built to test the influence of measured factors on the outcomes and to compensate for potential clustering of data. Data analysis including multilevel modeling will be conducted in collaboration with a biostatistician.

Schedule of investigational events

1. Screening and identification of subjects.
2. Baseline clinical examination of implants selected for the study. Case presentation and reinforcement of self-performed plaque control. Assessment of PROM. Professional mechanical infection control.
3. Radiographic examination prior to surgical therapy (within 4 weeks).
4. Surgical therapy including test and control treatment procedures at study sites.
5. 2 weeks - suture removal. Assessment of PROM.
6. 6 weeks - professional supra-mucosal cleaning and reinforcement of oral hygiene.
7. 6 months - clinical examination.
8. 12 months - clinical and radiological examination. Assessment of PROM.
9. 24 months - clinical examination.
10. 36 months - clinical and radiological examination. Assessment of PROM.
11. 48 months - clinical examination.
12. 60 months - clinical and radiological examination. Assessment of PROM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ≥1 implant (≥1 year of function) presenting with PPD ≥7 mm and BoP/Pus.
* Confirmed bone loss ≥3 mm at same implant(s)

Exclusion Criteria:

* Treated for peri-implantitis during previous 6 months
* Intake of systemic or local antibiotics during previous 6 months
* Systemic conditions affecting peri-implant tissues
* Systemic conditions impeding surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Treatment success (year 1) | Assessed at year 1
  Absence of bleeding/suppuration on probing, probing depth ≤5 mm and ≤1 mm recession of mucosal margin
Treatment success (year 3) | Assessed at year 3
  Absence of bleeding/suppuration on probing, probing depth ≤5 mm and ≤1 mm recession of mucosal margin
Treatment success (year 5) | Assessed at year 5
  Absence of bleeding/suppuration on probing, probing depth ≤5 mm and ≤1 mm

SECONDARY OUTCOMES:
Radiographic outcomes | Assessed at 1, 3 and 5 years
  Defect fill and crestal bone support
Patient-reported outcomes | Prior to intervention and at 1, 3 and 5 years
  Patient-reported outcomes assessed by questionnaire and in relation to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, Professor, Principal Investigator — Göteborg University
Locations (1):
- Department of Periodontology, Institute of Odontology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albouy JP, Abrahamsson I, Persson LG, Berglundh T. Implant surface characteristics influence the outcome of treatment of peri-implantitis: an experimental study in dogs. J Clin Periodontol. 2011 Jan;38(1):58-64. doi: 10.1111/j.1600-051X.2010.01631.x. Epub 2010 Nov 24. PMID 21092053
- [Background] Carcuac O, Abrahamsson I, Charalampakis G, Berglundh T. The effect of the local use of chlorhexidine in surgical treatment of experimental peri-implantitis in dogs. J Clin Periodontol. 2015 Feb;42(2):196-203. doi: 10.1111/jcpe.12332. Epub 2015 Jan 20. PMID 25385434
- [Background] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807
- [Background] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Background] Jepsen K, Jepsen S, Laine ML, Anssari Moin D, Pilloni A, Zeza B, Sanz M, Ortiz-Vigon A, Roos-Jansaker AM, Renvert S. Reconstruction of Peri-implant Osseous Defects: A Multicenter Randomized Trial. J Dent Res. 2016 Jan;95(1):58-66. doi: 10.1177/0022034515610056. Epub 2015 Oct 8. PMID 26450511
- [Background] Khoshkam V, Chan HL, Lin GH, MacEachern MP, Monje A, Suarez F, Giannobile WV, Wang HL. Reconstructive procedures for treating peri-implantitis: a systematic review. J Dent Res. 2013 Dec;92(12 Suppl):131S-8S. doi: 10.1177/0022034513509279. Epub 2013 Oct 24. PMID 24158331
- [Background] Roccuzzo M, Gaudioso L, Lungo M, Dalmasso P. Surgical therapy of single peri-implantitis intrabony defects, by means of deproteinized bovine bone mineral with 10% collagen. J Clin Periodontol. 2016 Mar;43(3):311-8. doi: 10.1111/jcpe.12516. Epub 2016 Mar 9. PMID 26800389
- [Background] Wohlfahrt JC, Lyngstadaas SP, Ronold HJ, Saxegaard E, Ellingsen JE, Karlsson S, Aass AM. Porous titanium granules in the surgical treatment of peri-implant osseous defects: a randomized clinical trial. Int J Oral Maxillofac Implants. 2012 Mar-Apr;27(2):401-10. PMID 22442781